CLINICAL TRIAL: NCT02807272
Title: A Phase 2 Study of Tipifarnib in Subjects With Chronic Myelomonocytic Leukemia, Other Myelodysplastic /Myeloproliferative Neoplasias, and Acute Myeloid Leukemia
Brief Title: Tipifarnib in Subjects With Chronic Myelomonocytic Leukemia, Other MDS/MPN, and Acute Myeloid Leukemia
Acronym: CMML/AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KO-TIP-004
Record Dates: First submitted 2016-06-15; First posted 2016-06-21 (Estimated); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Leukemia, Myelomonocytic, Chronic
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tipifarnib, Oral (Experimental): Single arm
  Interventions: Drug: Tipifarnib

INTERVENTIONS:
Drug: Tipifarnib — Oral tablet
  Other Names: R115777; Zarnestra

SUMMARY:
A Phase 2 study to investigate the antitumor activity in terms of overall response rate (ORR) of tipifarnib in approximately 36 eligible subjects with Myelodysplastic/Myeloproliferative Neoplasias (MDS/MPN), including Chronic Myelomonocytic Leukemia (CMML), and 36 eligible subjects with Acute Myeloid Leukemia (AML). Subjects received tipifarnib 1200 mg to be taken orally with food, twice daily, for 7 days in alternating weeks (Days 1 to 7 and Days 15 to 21) in 28-day cycles. Following amendment 3 subjects (Cohorts 1-4) will receive tipifarnib administered at a dose of 400 mg, orally with food, twice a day (bid) for 21 days in 28-day cycles.

DETAILED DESCRIPTION:
This Phase 2 study will investigate the antitumor activity in terms of ORR of tipifarnib in subjects with Myelodysplastic/Myeloproliferative Neoplasias (MDS/MPN cohorts) and Acute Myeloid Leukemia (AML cohorts). For MDS/MPN cohorts, this study will assess the antitumor activity of tipifarnib, in terms of ORR, in subjects with MDS/MPN, including CMML, who have a high ratio of expression of CXCR4 to CXCR2 (CXCR4/2 ratio) in their bone marrow and in those with a low CXCR4/2 ratio. For AML cohorts, this study will assess the antitumor activity of tipifarnib, in terms of ORR, in subjects with AML who have a high ratio of expression of CXCR4 to CXCR2 (CXCR4/2 ratio) in their bone marrow and in those with low CXCR4/2 ratio. Subjects enrolled in the study will consist of patients with KRAS, NRAS wild type status.

1. Subjects with MDS/MPN with high CXCR4/2 ratio
2. Subjects with MDS/MPN with low CXCR4/2 ratio
3. Subjects with AML with high CXCR4/2 ratio
4. Subjects with AML with low CXCR4/2 ratio

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age.
2. For subjects to be enrolled in the CMML or MDS/MPN cohorts:

   a. Diagnosis of CMML or MDS/MPN as defined by the World Health Organization (WHO) criteria (2008).
3. For subjects enrolled in the AML cohort:

   1. Documented pathological evidence of AML, as defined by WHO criteria (2008)
   2. Refractory to previous induction chemotherapy, relapsed disease, or age ≥ 60 and not appropriate for standard cytotoxic therapy due to age, performance status, and/or adverse risk factors according to the treating physician
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2.
5. Subject is willing and able to comply with scheduled visits, treatment plans, laboratory tests and other procedures (including bone marrow assessments).
6. At least 1 week since the last systemic therapy regimen prior to Cycle 1 Day 1. Subjects on a stable dose of hydroxyurea for at least 2 weeks prior to Cycle 1 Day 1 may continue on hydroxyurea until Cycle 1 Day 14. Subjects must have recovered to NCI CTCAE v. 4.03 < Grade 2 from all acute toxicities (excluding Grade 2 toxicities that are not considered a safety risk by the Sponsor and Investigator) or toxicity must be deemed irreversible by the Investigator.
7. Acceptable liver function:

   1. Total bilirubin ≤ upper limit of normal (ULN).
   2. AST (SGOT) and ALT (SGPT) ≤ 1.5 x ULN.
8. Acceptable renal function with serum creatinine ≤ 1.5 x ULN or a calculated creatinine clearance ≥ 60 mL/min using the Cockcroft-Gault or Modification of Diet in Renal Disease formulas.
9. Female subjects must be:

   1. Of non-child-bearing potential (surgically sterilized or at least 2 years post-menopausal); or
   2. If of child-bearing potential, subject must use a highly effective method of contraception, such as combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence. Both females and male subjects with female partners of child-bearing potential must agree to use a highly effective method of contraception for 2 weeks prior to screening, during, and at least 28 days after last dose of trial medication for females and 90 days for males. Female subjects must have a negative serum or urine pregnancy test within 72 hours prior to start of trial medication.
   3. And, not breast feeding at any time during the study.
10. Written and voluntary informed consent understood, signed and dated.

Exclusion Criteria:

1. Neoplasia harbours RAS mutation (NRAS mutant, KRAS mutant or double mutant)
2. Acute promyelocytic leukemia or Bcr-Abl positive leukemia (chronic myelogenous leukemia in blast crisis)
3. Clinically active CNS leukemia
4. CMML with t(5;12) that have not yet received imatinib.
5. Participation in any interventional study within 1 week of randomization or 5 half-lives of the prior treatment agent (whichever is longer).
6. Ongoing treatment with an anticancer agent for CMML, MDS/MPN or AML not contemplated in this protocol. Subjects on a stable dose of hydroxyurea for at least 2 weeks prior to Cycle 1 Day 1 may continue on hydroxyurea until Cycle 1 Day 14.
7. Hematopoietic stem cell transplantation (HSCT) performed within 3 months prior to Cycle 1 Day 1.
8. Concurrent use of granulocyte macrophage colony-stimulating factor (GM-CSF).
9. Prior treatment (at least 1 full treatment cycle) with a farnesyltransferase inhibitor.
10. Active coronary artery disease requiring treatment, myocardial infarction within the prior year, New York Heart Association grade III or greater congestive heart failure, cerebro-vascular attack within the prior year, or current serious cardiac arrhythmia requiring medication except atrial fibrillation.
11. Major surgery, other than diagnostic surgery, within 2 weeks prior to Cycle 1 Day 1, without complete recovery.
12. Active, concurrent malignancy requiring radiation, chemotherapy, or immunotherapy (excluding non-melanoma skin cancer, adjuvant hormonal therapy for breast cancer and hormonal treatment for castration sensitive prostate cancer).
13. Active and uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy. Known infection with human immunodeficiency virus (HIV), or an active infection with hepatitis B or hepatitis C.
14. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.
15. The subject has legal incapacity or limited legal capacity.
16. Significantly altered mental status that would limit the understanding or rendering of informed consent and compliance with the requirements of this protocol. Unwillingness or inability to comply with the study protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: TBD TBD, TBD, Principal Investigator
Locations (8):
- United States (8):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Weill Cornell Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants affected by chronic myelomonocytic leukemia (CMML) and myelodysplastic syndromes (MDS)/myeloproliferative neoplasms (MPN) were recruited across 10 sites in the United States between January 2017 and November 2020.
Pre-assignment Details: Participants w/ CMML were grouped by KRAS/NRAS status (wild type [WT], mutation [Mut], missing) & received tipifarnib 1200mg twice daily (BID) for 7 days, alternating weeks (Days 1-7, 15-21) in 28-day cycles. Following PA3 participants received tipifarnib 400mg orally w/ food, BID for 21 days in 28-day cycles. Those w/ MDS/MPN were stratified by ratio of expression (high/low) between CXCR4 & CXCR2 (CXCR4/2 ratio) receptors to receive tipifarnib 400mg orally, BID on Day 1-21 of each 28-day cycle.
Groups:
- KRAS/NRAS WT; KRAS/NRAS Mut; KRAS/NRAS Missing: Participants with CMML received tipifarnib at a starting dose of 1200 mg, BID, for 7 days in alternating weeks (Days 1 to 7 and Days 15 to 21) in 28-day cycles.
- CXCR4/2 High; CXCR4/2 Low: Participants with MDS/MPN received tipifarnib at a starting dose of 400 mg, orally, BID on Day 1 through 21 of each 28-day treatment cycle.
Period: Overall Study
Arm/Group | KRAS/NRAS WT | KRAS/NRAS Mut | KRAS/NRAS Missing | CXCR4/2 High | CXCR4/2 Low
Started | 23 | 12 | 2 | 3 | 4
Completed | 3 | 4 | 0 | 0 | 0
Not Completed | 20 | 8 | 2 | 3 | 4
Not completed — Death | 9 | 5 | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Permanent Withdrawal of Consent | 8 | 2 | 0 | 2 | 1
Not completed — Protocol-defined Disease Progression | 0 | 1 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 1 | 0 | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All enrolled participants who received at least one dose of tipifarnib.
Groups:
- Total: Total of all reporting groups
Arm/Group | KRAS/NRAS WT | KRAS/NRAS Mut | KRAS/NRAS Missing | CXCR4/2 High | CXCR4/2 Low | Total
Number analyzed (Participants) | 23 | 12 | 2 | 3 | 4 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (6.62) | 69.7 (6.68) | 76.0 (2.83) | 67.3 (2.89) | 70.5 (4.04) | 70.1 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 3 | 1 | 2 | 2 | 19
  Male | 12 | 9 | 1 | 1 | 2 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 12 | 2 | 3 | 3 | 41
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 10 | 1 | 3 | 4 | 38
  Black or African American | 2 | 0 | 1 | 0 | 0 | 3
  Native Hawaiian/other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 0 | 2
  American Indian/Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Other | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The ORR was estimated based on the number of participants who achieved an objective response (OR) (complete response [CR], complete cytogenetic remission [CCR], partial remission [PR], marrow response [MR], or clinical benefit [CB] performed by Principal Investigator according to the MDS/MPN International Working Group [IWG] criteria).
Time Frame: Up to 12 months
Population: Per Protocol Analysis Set (PP Analysis Set): Included participants who received at least 1 dose of tipifarnib and had a baseline disease assessment and at least 1 postbaseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | KRAS/NRAS WT | KRAS/NRAS Mut | KRAS/NRAS Missing | CXCR4/2 High | CXCR4/2 Low
Number analyzed (Participants) | 21 | 9 | 2 | 1 | 3
Participants
  CR | 0 | 0 | 0 | 0 | 0
  CCR | 0 | 1 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 1
  MR | 2 | 1 | 0 | 0 | 0
  CB | 1 | 1 | 1 | 0 | 0
  ORR | 3 | 3 | 1 | 0 | 1

2. Secondary Outcome: Duration of Response (DoR)
Description: DoR was measured from the date the participant first met the criteria of an OR to the date that the participant progressed or until death from any cause during the period of disease assessments. Participants without progression or death were censored at the date of the last disease assessment. Participants who received subsequent anticancer therapy were censored at the date of last disease assessment before subsequent anticancer therapy. The median duration of response and corresponding 95% CI was estimated using the Kaplan Meier method.
Time Frame: Up to approximately 15 months
Population: PP Analysis Set: Included participants who received at least 1 dose of tipifarnib and had a baseline disease assessment and at least 1 postbaseline disease assessment. Only participants who met the criteria for an OR and progressed or died were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | KRAS/NRAS WT | KRAS/NRAS Mut | KRAS/NRAS Missing | CXCR4/2 High | CXCR4/2 Low
Number analyzed (Participants) | 3 | 3 | 1 | 0 | 1
months | 14.6 [2.3 to NA] — Upper CI not calculable due to insufficient number of events. | NA [1.9 to NA] — Median and upper CI not calculable due to insufficient number of events. | 4.7 [NA to NA] — Upper and lower CI not calculable due to insufficient number of events. |  | NA [NA to NA] — Median and CI not calculable due to insufficient number of events.

3. Secondary Outcome: Progression Free Survival (PFS)
Description: The PFS time was defined as the time from the date of consent signed to the date of documented disease progression or death due to any cause, whichever occurred first. Participants without progression or death were censored at the date of the last disease assessment. Participants who received subsequent anticancer therapy were censored at the date of the last disease assessment before subsequent anticancer therapy. The Kaplan-Meier product-limit method was used to estimate the 1-year PFS rate, as well as the corresponding 95% CI.
Time Frame: 1 year
Population: PP Analysis Set: Included participants who received at least 1 dose of tipifarnib and had a baseline disease assessment and at least 1 post-baseline disease assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | KRAS/NRAS WT | KRAS/NRAS Mut | KRAS/NRAS Missing | CXCR4/2 High | CXCR4/2 Low
Number analyzed (Participants) | 21 | 9 | 2 | 1 | 3
months | 9.2 [3.6 to 12.9] | 4.1 [2.1 to NA] — Upper CI not calculable due to insufficient number of events. | 10.0 [NA to NA] — Upper and lower CI not calculable due to insufficient number of events. | NA [NA to NA] — Median and CI not calculable due to insufficient number of events. | 11.0 [1.7 to NA] — Upper CI not calculable due to insufficient number of events.

4. Secondary Outcome: Overall Survival (OS)
Description: OS time was defined as the time from the date of consent signed to the date of death due to any cause. Participants who were alive or lost to follow-up by the end of the study were censored at the date last known to be alive. The Kaplan-Meier method was used to estimate the proportion (%) of subjects without an event at 12 months, as well as their corresponding 95% CI.
Time Frame: Up to approximately 15 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | KRAS/NRAS WT | KRAS/NRAS Mut | KRAS/NRAS Missing | CXCR4/2 High | CXCR4/2 Low
Number analyzed (Participants) | 21 | 9 | 2 | 1 | 3
months | 14.4 [10.8 to NA] — Upper CI not calculable due to insufficient number of events. | NA [2.6 to NA] — Median and upper CI not calculable due to insufficient number of events. | 10.6 [6.9 to NA] — Upper CI not calculable due to insufficient number of events. | NA [NA to NA] — Median and CI not calculable due to insufficient number of events. | NA [11.0 to NA] — Median and upper CI not calculable due to insufficient number of events.

5. Secondary Outcome: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with it. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AE severity was rated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03.: grade 1(mild), grade 2(moderate), grade 3(severe), grade 4(life-threatening), grade 5(death). An AE was considered serious if resulted in any of the following: death, life-threatening, caused inpatient hospitalization or prolonged it, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, a congenital abnormality/birth defect, or was an important medical event.
Time Frame: Up to approximately 3 years
Population: FAS: All enrolled participants who received at least one dose of tipifarnib. Data was pooled into CMML and MDS/MPN arms as pre-specified in statistical analysis plan (SAP).
Measure: Count of Participants; unit: Participants
Groups:
- CMML: Participants with CMML were grouped by KRAS/NRAS mutational status (wild type [WT], mutation [Mut], missing) and given tipifarnib 1200mg twice daily (BID) for 7 days in alternating weeks (Days 1-7, 15-21) in 28-day cycles.
- MDS/MPN: Participants with MDS/MPN were stratified by ratio of expression (high or low) between CXCR4 and CXCR2 (CXCR4/2 ratio) receptors to receive tipifarnib at a dose of 400 mg, orally, BID on Day 1 through 21 of each 28-day treatment cycle.
Arm/Group | CMML | MDS/MPN
Number analyzed (Participants) | 37 | 7
Participants
  Any TEAE | 37 | 7
  Any tipifarnib-related TEAE | 37 | 6
  Any serious TEAE | 23 | 1
  Any tipifarnib-related serious TEAE | 13 | 1

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years
Description: FAS: All enrolled participants who received at least one dose of tipifarnib. Data was pooled into CMML and MDS/MPN arms as pre-specified in SAP.
Groups:
- MDS/MPS: Participants with MDS/MPN were stratified by ratio of expression (high or low) between CXCR4 and CXCR2 (CXCR4/2 ratio) receptors to receive tipifarnib at a dose of 400 mg, orally, BID on Day 1 through 21 of each 28-day treatment cycle.
Arm/Group | CMML | MDS/MPS
All-Cause Mortality (participants affected / at risk) | 17/37 | 1/7
Serious Adverse Events (participants affected / at risk) | 23/37 | 1/7
Other Adverse Events (participants affected / at risk) | 37/37 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CMML (N=37) | MDS/MPS (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Scrotal infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 3 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CMML (N=37) | MDS/MPS (N=7)
Anaemia (Blood and lymphatic system disorders) | 25 | 4
Leukocytosis (Blood and lymphatic system disorders) | 3 | 1
Sinus tachycardia (Cardiac disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 22 | 6
Diarrhoea (Gastrointestinal disorders) | 22 | 3
Constipation (Gastrointestinal disorders) | 13 | 2
Vomiting (Gastrointestinal disorders) | 10 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Dry mouth (Gastrointestinal disorders) | 4 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 4 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 23 | 4
Pyrexia (General disorders) | 8 | 1
Oedema peripheral (General disorders) | 8 | 0
Asthenia (General disorders) | 4 | 0
Chills (General disorders) | 4 | 0
Cellulitis (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 6 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 1
Platelet count decreased (Investigations) | 25 | 3
Blood creatinine increased (Investigations) | 16 | 2
Neutrophil count decreased (Investigations) | 15 | 2
White blood cell count decreased (Investigations) | 9 | 3
Lymphocyte count decreased (Investigations) | 5 | 3
Weight decreased (Investigations) | 5 | 0
Blood bilirubin increased (Investigations) | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 19 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 12 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Dizziness (Nervous system disorders) | 8 | 1
Headache (Nervous system disorders) | 7 | 2
Dysgeusia (Nervous system disorders) | 3 | 1
Memory impairment (Nervous system disorders) | 3 | 0
Paraesthesia (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 6 | 0
Anxiety (Psychiatric disorders) | 4 | 1
Confusional state (Psychiatric disorders) | 5 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 0
Renal cyst (Renal and urinary disorders) | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 0
Hypertension (Vascular disorders) | 6 | 0
Hypotension (Vascular disorders) | 5 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 0
Retching (Gastrointestinal disorders) | 1 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 2 | 0
Malaise (General disorders) | 2 | 0
Early satiety (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Corona virus infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0
International normalised ratio increased (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Haematoma (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are agreements in place between clinical trial sites and the Sponsor (or its agents) that govern discussion or publication of trial results by the sites or their employees after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT02807272/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT02807272/SAP_001.pdf